CLINICAL TRIAL: NCT05150405
Title: An Open, Dose-escalating Phase Ia Clinical Study to Evaluate the Tolerability, Safety, Pharmacokinetics and Preliminary Antitumor Activity of QLF31907 Injection in Patients With Advanced Cancer
Brief Title: A Phase Ia Clinical Study of QLF31907 Injection in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLF31907-101
Record Dates: First submitted 2021-10-28; First posted 2021-12-09 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLF31907 (Experimental): single arm with QLF31907 treatment
  Interventions: Drug: QLF31907

INTERVENTIONS:
Drug: QLF31907 — In this study, seven dose groups were proposed. The frequency of administration was once every two weeks, and four weeks was one therapeutic cycle. The subjects will receive six cycles of QLF31907 treatment at most.

SUMMARY:
This study is designed to evaluate the safety and tolerability of QLF31907 injection, to identify the maximum tolerated dose (MTD) and dose-limiting toxicity(DLT), and determine the recommended phase Ib dose(RPIbD) and recommended phase II dose (RP2D)in patients with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participated and signed a written informed consent form
2. Age ≥ 18 years, male or female
3. ECOG performance status of 0 or 1
4. Expected life-expectancy of more than 3 months
5. Solid tumors:

   Patients with histologically diagnosed head and neck squamous cell carcinoma (HNSCC), esophageal cancer (EC), renal cancer (RCC), melanoma, cervical cancer (CC), non-oncogene driver NSCLC and other solid tumors (requiring MSI-H/ dMMR signature gene) that are locally advanced, recurrent or metastatic that have failed or are intolerant to standard therapy.

   Hematologic tumors: patients with histologically diagnosed mediastinal large B-cell lymphoma (PMBCL), diffuse large B-cell lymphoma (DLBCL), mesenchymal large cell lymphoma (ALCL), peripheral T-cell lymphoma (PTCL), NKT-cell lymphoma, and high-grade B-cell lymphoma (R/R HGBL) that are intolerant or relapsed/refractory to standard therapy.
6. Patients with solid tumors have at least 1 measurable lesion according to RECIST v1.1. Patients with lymphoma have at least 1 measurable lesion or hypermetabolic lesion with 18F-FDG (18F-fluorodeoxyglucose) uptake according to Lugano2014 evaluation criteria.
7. Adequate organ function prior to first use of the trail drug (no blood components, cell growth factors, leukocyte-raising drugs, platelet-raising drugs, etc., or hepatoprotective therapy is allowed within 14 days prior to obtaining laboratory tests)

   1. Absolute neutrophil count ≥ 1.5 x 109/L
   2. Platelet count ≥ 80 × 109/L (≥ 90 × 109/L in patients with hepatocellular carcinoma)
   3. Hemoglobin ≥ 90g/L
   4. Serum creatinine ≤ 1.5 × upper limit of normal (ULN); for patients with creatinine level > 1.5 × ULN, according to Cockcroft-Gault formula for creatinine clearance (CLcr) ≥ 60 mL / min
   5. Total bilirubin ≤ 1.5 × ULN
   6. AST and ALT ≤ 2.5 × ULN (for Gilbert's syndrome, hepatocellular carcinoma or the presence of liver metastases, ≤ 5 × ULN)
   7. Coagulation function: prothrombin time ≤ 1.5 × ULN, activated partial thromboplastin time ≤ 1.5 × ULN, international normalized ratio ≤ 1.5 × ULN
   8. Cardiac left ventricular ejection fraction (LVEF) > 50%
8. Subjects (both female and male) agree to use effective contraception from the time they sign the informed consent form until 180 days after the last use of the trial drug.
9. Recovery from all the other reversible AEs from prior antineoplastic therapy prior to the first administration of the trail drug (i.e. ≤ grade 1, according to CTCAE v5.0), excluding alopecia (any grade) and ≤ grade 2 peripheral sensory neuropathy or lymphocytopenia. Subjects who develop other abnormalities without clinically significant or investigator-judged risk-free toxicity will be enrolled only after discussion and approval by the sponsor and investigator.

Exclusion Criteria:

1. Previous treatment with 4-1BB agonist or 4-1BB recombinant fusion protein
2. Received antitumor therapy with chemotherapy, biologic therapy, endocrine therapy, immunotherapy, or monoclonal antibodies within 4 weeks prior to the first use of the trail drug, with special circumstances as follows.

   1. Including those who have received oral fluorouracil analogues, small-molecule targeted drugs and herbal or Chinese patent medicine with antitumor indications within 2 weeks prior to the first use of the trail drug
   2. Including those who have received mitomycin or nitrosoureas within 6 weeks prior to the first use of the trail drug
   3. Including those who have received cell-based therapy or antitumor vaccine within 8 weeks prior to the first use of the trail drug
   4. In subjects with a high tumor burden, treatment to reduce tumor burden for the purpose of preventing tumor lysis syndrome during the course of the trial is excluded
3. Subjects with central nervous system (CNS) metastases or clinical manifestations of CNS involvement, soft meningeal metastases, or spinal cord compression due to metastases prior to signing informed consent. Except for symptomatic CNS metastases that have been treated and stable for ≥4 weeks prior to the first administration of the investigational drug and who have been off systemic hormone (at any dose) therapy for >2 weeks.
4. Subjects with uncontrolled exudate or leaky fluid (thoracic, pericardial, or abdominal) or one of thoracic fluid >500 ml, pericardial fluid >100 ml, or abdominal fluid ≥1000 ml
5. History of autoimmune disease (including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism [except for subjects who can be controlled by hormone replacement therapy only]; except for subjects with skin diseases that do not require systemic treatment such as vitiligo, psoriasis and alopecia areata; except for type I diabetes or asthma that has completely resolved in childhood and does not require any intervention in adulthood, such as asthma patients who require medical intervention with bronchodilators are not included)
6. Have had other active malignancies within 3 years prior to study entry (from the time of signing informed consent form). Cured basal or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, intraductal carcinoma in situ of the breast and papillary thyroid cancer were excluded
7. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis (hepatitis B: defined as positive hepatitis B virus surface antigen [HBsAg] and e antigen [HBeAg] test results, or HBV-DNA ≥ 20 IU/ml, or HBV-DNA ≥ 1000 copies/ml, or persistent liver function abnormal, or tissue biopsy with hepatitis pathology, or cirrhosis; hepatitis C: defined as positive hepatitis C antibody [HCV-Ab] and HCV-RNA above the lower limit of detection of the analytical method), combined hepatitis B and C co-infection; syphilis spirochete infection; Mycobacterium tuberculosis infection
8. History of hepatitis (non-alcoholic steatohepatitis, alcoholic or autoimmune hepatitis) and cirrhosis
9. Subjects with the following cardiovascular events including but not limited to: myocardial infarction, severe/unstable angina, NYHA class 2 or higher cardiac insufficiency and clinically significant supraventricular or ventricular arrhythmias, prolonged QT interval and need for clinical intervention within 6 months prior to study entry (from the time of signing informed consent form); congenital heart disease such as clinically significant heart valve stenosis, insufficiency of closure and cardiomyopathy
10. Systemic antibiotic use for ≥ 7 days within 4 weeks prior to first dose, or unexplained fever > 38.5°C during screening/prior to first dose (fever due to oncologic causes may be enrolled, as determined by the investigator)
11. Subjects with a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation/history of bone marrow transplantation treatment, autologous stem cell transplantation within 180 days
12. Participation in any other drug clinical study within 4 weeks prior to the first dose and use of other study drugs (except minerals, vitamins), or no more than 2 weeks from the last study drug (half-life ≤ 3 days) and no more than 28 days from the last study drug (half-life > 3 days)
13. Subjects with a known history of psychotropic substance abuse, alcohol or drug abuse; a clear previous history of neurological or psychiatric disorders, including epilepsy or dementia.
14. Known hypersensitivity to the study drug or any of its excipients; or a history of severe allergic reactions to other monoclonal antibodies; or are allergic.
15. Women who are pregnant or breastfeeding, except for women who are breastfeeding and may stop breastfeeding during the study; patients who are intending or planning to have children during the study.
16. History of idiopathic pulmonary fibrosis, pneumoconiosis, asbestosis (including drug-induced lung injury)
17. Active pneumonic lesions detected on CT chest scan during the screening period
18. Systemic immunosuppressive therapy with drugs including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, and anti-TNFα (tumor necrosis factor) drugs, except for localized and short-term small doses use within 2 weeks of the first administration of trail drug
19. Subjects who have undergone local radiation therapy for palliation within 7 days prior to the first dose; subjects who have received radiation therapy with more than 30% of the bone marrow irradiated or whole brain radiation therapy within 4 weeks prior to the first dose
20. Combined second tumor requiring concurrent treatment with other antineoplastic agents (except hormonal therapy for breast and prostate cancer)
21. Presence of uncontrolled or poorly controlled underlying respiratory, circulatory and endocrine diseases such as chronic obstructive pulmonary disease, hypertension, coronary artery disease, diabetes mellitus and hyperthyroidism
22. Presence of other serious physical or mental illnesses or abnormal laboratory tests that may increase the risk of participation in the study or interfere with the results of the study, and subjects who are not suitable for participation in this study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 28 days
  The DLT of QLF31907 will be determined.
Maximum tolerated dose(MTD) | up to 2 years
  The MTD of QLF31907 will be determined.

SECONDARY OUTCOMES:
Frequency of adverse events of QLF31907 | up to 2 years
  Adverse events will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Cmax of QLF31907 | up to 2 years
  Peak Plasma Concentration (Cmax) of QLF31907 will be determined.
AUC of QLF31907 | up to 2 years
  Area under the plasma concentration versus time curve (AUC) of QLF31907 will be determined.
Tmax of QLF31907 | up to 2 years
  Time to Cmax (Tmax) of QLF31907 will be determined.
Immunogenicity of QLF31907 | up to 2 years
  Frequency of anti-drug antibodies (ADA) against QLF31907 will be determined.
Anti-tumor activity of QLF31907 | up to 2 years
  Solid tumor response will be determined by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1), and lymphoma response will be determined by criteria of lugano 2014.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China